CLINICAL TRIAL: NCT01346579
Title: PIK3CA Mutation Status as a Biomarker in Elderly Women With Breast Cancer
Brief Title: Biomarkers in Tissue Samples From Older Women With Breast Cancer
Status: Terminated | Type: Observational
Why Stopped: Study closed prematurely.
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-151101; CDR0000699810 (Registry Identifier: NCI Physician Data Query)
Record Dates: First submitted 2011-04-30; First posted 2011-05-03 (Estimated); Last update posted 2016-07-04 (Estimated); Status verified 2016-07

CONDITIONS: Breast Cancer
Keywords: stage IA breast cancer; stage IB breast cancer; estrogen receptor-positive breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tissue
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative sciences

SUMMARY:
This research trial studies phosphatidylinositol-4,5-bisphosphate 3-kinase, catalytic subunit alpha (PIK3CA) mutation analysis in tissue samples from older patients with stage I breast cancer. Studying samples of tissue from patients with stage I breast cancer in the laboratory may help doctors learn more about changes that occur in deoxyribonucleic acid (DNA) and identify biomarkers related to cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

To assess the relapse free-survival difference between patients with PIK3CA mutated and wild-type (WT) tumors and therefore validate PIK3CA mutation status as an important biomarker in women 70 years or older diagnosed with breast cancer.

OUTLINE:

Previously collected tissue samples are analyzed via mutation analysis of PIK3CA.

ELIGIBILITY:
* Participants with stage I breast cancer (T1N0M0) and estrogen-receptor status positive or unknown
* Patients underwent lumpectomy with negative margins and were clinically node-negative

Min Age: 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with breast cancer enrolled on Cancer and Leukemia Group B 9343
Sampling Method: Non-Probability Sample
Enrollment: 505 (Actual)
Dates: Start 2011-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Breast cancer-free interval for patients with PIK3CA-mutated tumors | baseline
Tumor size | baseline
Estrogen receptor status | baseline
Lymph node status | baseline
Treatment group associated with PIK3CA expression | baseline

SECONDARY OUTCOMES:
Overall survival associated with PIK3CA | baseline
Breast cancer specific survival associated with PIK3CA expression | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ellen Moynahan, MD, Study Chair — Memorial Sloan Kettering Cancer Center